CLINICAL TRIAL: NCT00046137
Title: Combined Use of Teriparatide and Raloxifene in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 6817; B3D-MC-GHCD
Record Dates: First submitted 2002-09-20; First posted 2002-09-23 (Estimated); Last update posted 2006-07-20 (Estimated); Status verified 2006-07

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Teriparatide; Raloxifene Hydrochloride

INTERVENTIONS:
Drug: teriparatide
Drug: raloxifene
Drug: placebo

SUMMARY:
The purpose of this study is to compare treatment with both teriparatide and raloxifene with teriparatide alone. The study will evaluate any side effects that may be associated with the two drugs and may help to determine whether teriparatide and raloxifene together can help patients with osteoporosis more than teriparatide alone.

ELIGIBILITY:
Inclusion Criteria

* Must be diagnosed with osteoporosis.
* Must be female, age 45 through 85.
* Must be at least 5 years postmenopausal.
* Must be free of other severe or chronically disabling conditions.
* Must be able to properly use injection device.

Exclusion Criteria

* Must not have bone diseases other than osteoporosis.
* Must not have history of certain cancers.
* Must not have certain medical diseases (inflammatory bowel disease, malabsorption syndrome, kidney or bladder stones, venous thrombi or emboli, recent vaginal bleeding due to unknown causes).
* Must not have taken or are currently taking certain types of medicines.
* Must not have known allergy to the study agent or SERM.

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician"., Anaheim, California
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician"., Oakland, California
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician"., Altamonte Springs, Florida
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician"., Chicago, Illinois
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician"., Cedar Rapids, Iowa
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician"., Baltimore, Maryland
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician"., Hagerstown, Maryland
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician"., Voorhees Township, New Jersey
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician"., Cleveland, Ohio
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician"., Oklahoma City, Oklahoma
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician"., Portland, Oregon
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician"., Duncansville, Pennsylvania
  - "For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician"., Dallas, Texas